# A One-Day ACT Workshop for Emotional Eating

**Study Protocol** 

Frayn & Knäuper

**September 16, 2018** 

#### Methodology/Procedures

- 1. **Recruitment:** Participants will be recruited through flyers placed on the university campus as well as office buildings and community locations such as local gyms and doctor's offices. Advertisements will also be placed in the university's staff newsletter.
- 2. Prescreening: To determine eligibility, interested individuals will be assigned an ID number and asked to complete the Dutch Eating Behavior Questionnaire Emotional Eating subscale (DEBQ-EE, van Strien et al., 1986) online through SurveyMonkey to see whether they are eligible. The questionnaire will also ask them their age to ensure that they are over 18, as we are only recruiting adults. All of those who meet criteria for emotional eating (score of 3.25 or higher on the emotional eating subscale) will be eligible to participate and will be contacted to schedule their participation in the workshop.
- 3. Baseline assessments: After they have consented to participate in the study, all participants will complete a demographics questionnaire, the DEBQ-EE, the Distress Tolerance Scale (DTS; Simons & Gaher, 2005), the Food Acceptance and Awareness Questionnaire (FAAQ; Juarascio, Forman, Timko, Butryn, & Goodwin, 2011), and the Mindful Eating Questionnaire (MEQ; Framson et al., 2009) prior to attending the workshop. They will also be asked a series of questions pertaining to values clarification and commitment in relation to emotional eating. Finally, they will be asked to complete two additional items recording the number of times they engaged in emotional eating as well as how much often they were able to stop emotional eating after starting. These items were developed by the authors. All questionnaires will be completed online through SurveyMonkey.

4. **Intervention:** Workshops will be 4-6 hours in length and held on Saturdays. They will be facilitated by clinical psychology PhD students. The intervention will be modeled after Frayn and Knäuper's (2016) brief emotional eating intervention, which was derived from Forman et al.'s (2013) "Mind Your Health program". During the workshop, the following topics will be discussed, based on the three processes of ACT relevant to emotional eating identified in Forman and Butryn's (2014) review:

# (1) Values Clarification and Commitment

- a. Exploring values and why it is important for participants to reduce their emotional eating. Values clarification will be emphasized to allow participants to identify that emotional eating is inconsistent with values pertaining to health and wellness. This values clarification will set the framework for motivating alternative, valueconsistent behaviours.
- b. Using values to make decisions and to engage in committed action (teaching the BOLD technique and walking participants through examples). Participants will be asked to brainstorm alternative, value-consistent behaviours that do not involve eating.

# (2) Acceptance/Distress Tolerance

- a. Introducing acceptance, specifically acceptance of negative emotions, within the ACT model (e.g., use tug-of-war metaphor and dropping the rope to elucidate this). Using acceptance in the context of emotional eating to explain that participants do not have to respond to their negative emotions by eating.
- b. Introducing the concept of urge surfing, allowing participants to normalize cravings that arise as a result of negative emotions. Teaching participants concrete

steps to employ urge surfing to sit with negative emotions and cravings, rather than acting on them by eating.

### (3) Mindfulness/Awareness

a. Introducing mindful eating. Participants will be asked to participate in an exercise where they are taught to mindfully eat dark chocolate. Mindful eating will be applied to emotional eating, as emotional eating is typically a mindless experience. Participants will be encouraged to pay mindful awareness of their hunger/satiety cues, and eat mindfully in a way that is physically and psychologically satisfying.

Following the introduction and application of these three techniques, a discussion will be held to review what was taught and to identify which techniques resonate most with participants. The facilitator will answer/clarify any questions people may have about any of the concepts taught. Towards the end of the workshop, the facilitator will also introduce the concept of habit formation and the importance of practicing the techniques such that they become automatic. The workshop will conclude with committed action, bringing the discussion back to the commitment to values discussed at beginning of session.

5. At the very end of the afternoon session, a brief discussion will be had to gain participants' insight on the program to qualitatively assess treatment acceptability.

Workshop facilitators will also be asked to provide their perceptions of how the workshop was received by participants. Qualitative discussion prompts will be based on recommendations by O'Cathain et al. (2015) for using qualitative data to inform feasibility studies. The contents of these discussions will be subject to thematic analysis to identify emergent themes pertaining to treatment acceptability.

6. **2-weeks and 3-month follow-ups:** At these time points, participants will be asked to complete the same battery of questionnaires they completed prior to taking the workshop. The purpose of these follow-up assessments is to assess changes in these variables from baseline to 2-weeks and 3-months post-intervention to examine the effectiveness of the workshop in the short and long term.

#### References

- Forman, E. M., & Butryn, M. L. (2014). A new look at the science of weight control: How acceptance and commitment strategies can address the challenge of self-regulation.

  Appetite, 84, 171-180.
- Forman, E. M., Butryn, M. L., Juarascio, A. S., Bradley, L. E., Lowe, M. R., Herbert, J. D., & Shaw, J. A. (2013). The mind your health project: A randomized controlled trial of an innovative behavioral treatment for obesity. *Obesity*, *21*, 1119-1126.
- Framson, C., Kristal, A. R., Schenk, J. M., Littman, A. J., Zeliadt, S., & Benitez, D. (2009).

  Development and validation of the mindful eating questionnaire. *Journal of the American Dietetic Association*, 109(8), 1439-1444.
- Frayn, M. & Knäuper, B. (2016). Weight loss program for emotional eaters: Physician manual and participant handouts. McGill University, Montreal.
- Juarascio, A., Forman, E., Timko, A., Butryn, M., & Goodwin, C. (2011). The development and validation of the food craving acceptance and action questionnaire (FAAQ). *Eating Behaviors*, 12, 182-187.
- O'Cathain, A., Hoddinott, P., Lewin, S., Thomas, K. J., Young, B., Adamson, J., Jansen, Y. J., Mills, N., Moore, G., & Donovan, J. L. (2015). Maximising the impact of qualitative research in feasibility studies for randomised controlled trials: Guidance for researchers. *Pilot and Feasibility Studies*, 7, 1-32.
- Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and validation of a self-report measure. *Motivation and Emotion*, *29*, 83-102.

van Strien, T., Frijters, J., Bergers, G., & Defares, P. B. (1986). The Dutch Eating Behavior Questionaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. *International Journal of Eating Disorders*, *5*, 295-315.